CLINICAL TRIAL: NCT06874452
Title: Pain, Anxiety and Anesthetic Satisfaction for Patient With Different State Anxiety Underwent Cataract Surgery With Topical Anesthesia. An Extension Test of Whether to Use Oral Anti-anxiety Drugs (XANAX) When Patients Choose Second Eye Cataract Surgery After Unblinding, and Analyze Their Anxiety, Satisfaction and Pain Satisfaction
Brief Title: An Extension Test of Whether to Use Oral Anti-anxiety Drugs (XANAX) When Patients Choose Second Eye Cataract Surgery After Unblinding, and Analyze Their Anxiety, Satisfaction and Pain Satisfaction
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202410134MINC
Record Dates: First submitted 2025-03-04; First posted 2025-03-13 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Ophthalmology; Cataract Surgery Anesthesia; Oral Anxiolytic; Satisfaction Survey
Keywords: oral anti-anxiety drugs; oral anxiolytic; ophthalmology; cataract surgery anesthesia; satisfaction survey
MeSH Terms: interventions — Alprazolam

STUDY DESIGN:
Intervention Model Description: open label, double-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xanax (Experimental): 0.5mg XANAX or 0.25MG XANAX for patients older than 65 years or with liver disease.
  Interventions: Drug: Xanax
- placebo (Placebo Comparator): The placebo tablet is visually identical to the experiment group.
  Interventions: Other: Placebo Tablets

INTERVENTIONS:
Drug: Xanax — The patients will each receive a single tablet of 0.5mg XANAX 30 minutes before surgery. Patients older than 65 years or with liver disease will receive a reduced dose of 0.25 mg rather than 0.5 mg of oral XANAX 30 minutes before surgery.
  Arms: Xanax
Other: Placebo Tablets — The patients will each receive a single tablet of placebo 30 minutes before surgery.
  Arms: placebo

SUMMARY:
Phacoemulsification is one of the most used surgical methods for cataract surgery today, and the surgeries are under the anesthetic and sedative to make it comfortable and safe for patients. The most important issue is which method is the best for reducing the patient's anxiety, pain, and discomfort during surgery. Previous studies have analyzed the impact of intravenous injection of sedative on the quality of phacoemulsification surgery; however, the impact of oral anti-anxiety drugs (XANAX) on cataract surgery has not been intensively studied. Therefore, the purpose of this study is to investigate the impact of XANAX on satisfaction in cataract surgery. Oral sedation is more convenient and safer than intravenous sedation. Therefore, the investigators will further analyze whether patients using oral anti-anxiety drugs will have an improvement in the pain, anxiety, overall satisfaction, and side effects related to nausea and dizziness in the phacoemulsification surgery. This study will detailed record the patient's status in various aspects using questionnaire scales and scores. Through this research, the investigators will have the opportunity to comprehensively improve the surgical quality of cataract patients in a safe and convenient manner. The investigators plan to collect data from patients who participated in the study "Anxiety and surgery satisfaction for cataract patient with different state anxiety" (Research Ethics Committee Case No.: 202302067MINB) from October 2023 to August 2025, and plan to undergo phacoemulsification and intraocular lens implantation surgery in their second eye with local anesthetic at the Department of Ophthalmology, National Taiwan University Hospital. The sample size of 250 participants was determined based on the type of intervention, expected effect size, outcome variability, desired statistical significance, trial power, and experiences from similar studies. Vulnerable populations and those with any relevant contraindications will be excluded during the enrollment process. All medical records and surgical process data, including privacy-related information, will only be accessible to professional medical personnel for analysis. The focus of this study will be on intraoperative satisfaction, pain scores, relevant discomfort symptoms during the surgery, and postoperative anxiety assessment scales.

DETAILED DESCRIPTION:
BACKGROUNDS Nowadays, phacoemulsification for cataract treatment is the most common surgical procedure performed and anesthetics procedure has been shifted from retrobulbar or peribulbar anesthesia to topical anesthesia (TA). Phacoemulsification under TA proved to be a safe and low risk procedure with the incidence of adverse events requiring medical emergency team interventions to be 0.04%. However, it is not uncommon that patients can suffer from pain, anxiety and unpleasant visual sensation during this procedure. Complementary sedation has long been thought to alleviate the anxiety and pain of the patient during surgery with local anesthesia. Studies revealed that approximately one fourth of the patients underwent phacoemulsification under TA or retrobulbar anesthesia requested additional intravenous sedation of midazolam. [8] However, the intravenous sedation, such as midazolam, propofol, or etomidate, increase the risk of additional anesthetic complications of heart rate, blood pressure, body temperature, and nausea, [9,10] and therefore, anesthesia monitoring was mandatory during the surgery.

Compared with intravenous sedation, oral sedation is less costly and less invasive. Studies with different oral sedation agents revealed different effects. In the study of 41 patients serving themselves as control, patients reported more pain and photophobia in the surgery with TA alone than the other with midazolam syrup and oral transmucosal fentanyl citrate. However, two studies comparing oral diazepam or triazolam with intravenous midazolam showed similar rates of anxiety and pain or noninferior satisfaction. Moreover, the randomized control trial containing 50 procedures in each groups revealed that patients received TA alone during phacoemulsification reported similar pain or anxiety level to those received complementary intravenous midazolam. Despite the abundant results from above, nearly 40% patients reported moderate to extremely anxiety during phacoemulsification under TA, and approximate 7% of patients rated themselves extreme anxiety or were diagnosed as anxiety. A simple comparison between with or without complementary sedation for general patients underwent phacoemulsification with TA is merely not enough. Further investigations to reduce the anxiety experienced during phacoemulsification with TA according to patients' characteristics is therefore mandatory. Previous studies had showed that patients with higher level of trait anxiety reported higher anxiety response for a stressful situation. Preoperative anxiety levels were also reported to be a significant predictor of pain experience during phacoemulsification with TA. The need for complementary sedation could be different in patients with different trait anxiety. Furthermore, different severity levels of anxiety and pain were experienced during the first and second eye surgery. Therefore, in this study, the investigators will investigate the trait anxiety of patients planned for phacoemulsification under TA and its effect on their anesthetic satisfaction with complementary oral sedation. The investigators will also analysis the anxiety and pain experienced in the first and second eye phacoemulsification in patients with different levels of trait anxiety. The investigators choose alprazolam as the oral sedative. It was reported to have a shorter half-life and less side effects of drowsiness and lightheadedness than diazepam used in previous studies.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years old.
2. Enrolled in "Anxiety and surgery satisfaction for cataract patient with different state anxiety" (Research Ethics Committee Case No.: 202302067MINB).
3. Plan to undergo phacoemulsification and intraocular lens implantation surgery with topical anesthetic on the second eye at the Department of Ophthalmology.
4. Subject who does not have side effect from XANAX.

Exclusion Criteria:

1. Presence of any surgery contraindications.
2. Presence of any medication contraindications.
3. Inability to provide clear and complete answers to relevant questionnaires, or expression of no preoperative anxiety during the outpatient visit, or scores below 21 on the STAI-S or STAI-T assessment.
4. Regular use of anti-anxiety medications, sleeping pills, or analgesics before the procedure.
5. Pregnancy or breastfeeding during the preoperative period.
6. Severe corneal diseases, overripe cataracts, small pupils, or lens dislocation leading to difficulties in conventional surgery.
7. Patients under surface anesthesia who cannot fully cooperate with the surgical procedure.
8. Pregnant or uncertain pregnancy status (women under 55 years old to be verbally asked by research team members).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Anesthesia Satisfaction Assessment | 1 day
  The anesthesia satisfaction rating scale evaluates patients' satisfaction with the anesthesia experience during surgical procedures, focusing on factors such as pain management, comfort, and communication with the anesthesia team. The scales typically use a numerical rating system, such as a 10-point scale, where higher scores indicate greater satisfaction.

SECONDARY OUTCOMES:
The change of preoperative and postoperative anxiety level | 1 day
  The change of preoperative and postoperative anxiety level is evaluation with State-Trait Anxiety Inventory (STAI) and Beck Anxiety Inventory (BAI). STAI is focus on state anxiety (SA) and trait anxiety (TA). The inventory comprises 40 items, with 20 items assessing state anxiety and 20 items assessing trait anxiety. Each item is rated on a 4-point scale (1 to 4), resulting in a total score range of 20 to 80 for both SA and TA. Higher scores indicate more severe anxiety. BAI consists of 21 items covering physiological and cognitive anxiety symptoms, such as palpitations, breathlessness, and tension. Each item is rated on a 4-point scale (0 to 3) based on the frequency or severity of symptoms, with a total score range of 0 to 63. Higher scores indicate more severe anxiety.
Level of postoperative pain | 1 day
  The immediate postoperative pain levels is documented to assess the patient's postoperative satisfaction. The pain level is rated on a 10-point scale (0 to 10). 0 point represents no pain, 1-2 points represent mild pain, 3-4 points represent moderate pain, 5-6 points represent severe pain, 7-8 points represent very severe pain, and 9-10 points represent worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: Chiun Ho Hou, Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No